CLINICAL TRIAL: NCT05934175
Title: Efficacy, Mechanisms of Change and Cost Effectiveness of Intensive Exposure-based Treatment for PTSD: a Randomized Controlled Trial
Brief Title: Intensive Treatment Versus Standard Weekly Prolonged Exposure for Adults With Post-Traumatic Stress Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Maria Bragesjo, Clinical psychologist, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-02329-01
Record Dates: First submitted 2023-06-26; First posted 2023-07-06 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD; intensive treatment; prolonged exposure; massed treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Prolonged exposure will be offered in a massed format with a total of nine 60 minutes sessions of imaginal exposure and processing and five 2 hour group session with psychoeducation, rationales and in vivo exposure during one treatment week followed by three individual 60 minutes sessions 1, 2 and 4 weeks afterwards.
Who Masked: Outcomes Assessor
Masking Description: Blinded assessors are used
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive treatment with prolonged exposure (Experimental): Intensive prolonged exposure delivered for five consecutive days comprising nine individual sessions and five group sessions followed by three individual session one, two and four weeks afterwards.
  Interventions: Behavioral: Intensive treatment with prolonged exposure
- Weekly delivered prolonged exposure (Active Comparator): 15 weekly delivered, individual prolonged exposure sessions (gold standard treatment)
  Interventions: Behavioral: Weekly delivered prolonged exposure

INTERVENTIONS:
Behavioral: Intensive treatment with prolonged exposure — Intensive treatment with prolonged exposure
  Arms: Intensive treatment with prolonged exposure
Behavioral: Weekly delivered prolonged exposure — Weekly delivered prolonged exposure sessions for 15 weeks
  Arms: Weekly delivered prolonged exposure

SUMMARY:
The goal of this clinical trial is to compare a novel, massed treatment format of prolonged exposure to gold standard trauma focused cognitive behavioral therapy (weekly delivered prolonged exposure) for post-traumatic stress disorder.

The objective with this study is to investigate efficacy, mechanisms of change and cost effectiveness of intensive prolonged exposure (I-PE) in regular Swedish psychiatric care.

Adult patients with post-traumatic stress disorder will be randomly assigned to receive either gold standard prolonged exposure weekly for 15 weeks or 5 days of intensive treatment with the addition of three booster sessions dispersed 1, 2 and 4 weeks after completion of the massed treatment period.

DETAILED DESCRIPTION:
PTSD is one of the most common psychiatric disorders and is strongly linked to subsequent psychiatric and medical problems. Trauma-focused cognitive behavioral therapy (CBT-T) such as prolonged exposure is an effective treatment for PTSD and is recommended in most clinical guidelines as first-line treatment. However, the treatment period often lasts 3-5 months, which is believed to be a contributing factor to the high dropout rate that has suggested to be a major factor to why a significant proportion of patients fail to demonstrate clinically significant symptom change. In response, more intensive treatment approaches i have been developed based on the notion that frequency of treatment sessions are a potential mechanism for retention. Preliminary research shows intensive trauma focused treatment (I-PE) to be as effective as when the treatment is delivered by weekly sessions, but with the advantage that the recovery rate is faster and the proportion of patients who drop out decreases.

Before this type of treatment can be offered in regular care in Sweden, it needs to be further evaluated. If I-PE would be found to effective, this project has the potential to be the first step towards implementation of a novel, superior and more cost-effective mode of treatment delivery for adults with PTSD in regular Swedish health care. The intensive treatment format has yet to be directly compared to gold-standard CBT-T, and that is what we propose to do in this trial.

The study is a single-blind, parallel-group superiority randomized controlled trial with 140 patients (70 per arm) will compare intensive prolonged exposure to gold standard weekly delivered prolonged exposure. The primary outcome is the blind-rater administered Clinician-Administered PTSD Scale for DSM-5 (CAPS-5).

Secondary outcomes are cost effectiveness, speed of response, response and remission rates, dropout rate, and negative effects. The investigators hypothesis that participants in the massed treatment format will improve faster than patients that receive weekly sessions, but for the rest of the secondary outcomes, the investigators have no directed hypotheses.

The trial will also be preregistered at the Open Science Framework.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or above,
* Primary PTSD diagnosis
* Fluent in Swedish
* Sign informed consent
* Able to attend either I-PE or 15 weekly sessions of PE

Exclusion Criteria:

* Initiation or adjustment of any psychotropic medication within the last 4 weeks prior to commencement of treatment
* Serious mental health symptoms, such as mania, psychosis, alcohol, or substance use disorders or current suicide risk warranting immediate clinical attention
* Ongoing evidence-based trauma-focused psychological treatment
* Ongoing trauma-related threat (e.g. living with a violent spouse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptoms as assessed by the Clinician Administered PTSD Scale (CAPS-5) | Baseline, 1-month (primary endpoint), 6-month and 12-month post-treatment
  The CAPS-5 is structured interview that assesses the Diagnostic and Statistical Manual of Mental Disorders version 5 (DSM-5) criteria for PTSD (Weathers et al., 2013). Each item is rated on a severity scale ranging from 0 (Absent) to 4 (Extreme/incapacitating) and combines information about frequency and intensity for each of the 20 symptoms. Total Score (Range 0-80 with higher scores representing more PTSD symptoms.

SECONDARY OUTCOMES:
Change in PTSD symptoms as assessed by the PTSD Check List - DSM-5 (PCL-5) | Baseline, through the treatment period up to 15 weeks after inclusion and at 1-month, 6-month and 12-month post-treatment
  The PCL-5 is a 20-item self-report measure based upon the Diagnostic and Statistical Manual (DSM-5) criteria for PTSD. Total Score (Range 0-80 with higher scores representing more PTSD symptoms.
Change in ICD-11 PTSD and complex PTSD symptoms as assessed by the International Trauma Questionnaire (ITQ). | Baseline, through the treatment period and 1-month, 6-month and 12-month post-treatment
  The ITQ includes six items measuring each PTSD symptom cluster and these items measure how bothersome each symptom has been in the past month. The ITQ also includes six items measuring each 'Disturbance in Self-Organization' (DSO) symptom in complex PTSD. These items measure how a respondent typically feels, thinks about oneself, and relates to others. The PTSD and DSO symptoms are accompanied by three items measuring associated functional impairments in the domains of social, occupation, and other important areas of life. All items are answered on a 5-point Likert scale ranging from 0 (Not at all) to 4 (Extremely). Thus, PTSD and DSO symptom scores range from 0 to 24 and CPTSD symptom scores range from 0 to 48. Higher scores represents more PTSD and complex PTSD symptoms.
Change in depressive symptoms as measured by the Patient Health Questionnaire-9 (PHQ-9) | Baseline, immediately after treatment completion, 1-month, 6-month and 12-month post-treatment
  The PHQ-9 is a widely used and well-validated instrument for measuring the severity of depressive symptoms. Scores are calculated based on how frequently a person experiences 9 symptoms of depression ranging from "not at all" response is scored as 0; "several days" response is 1; "more than half the days" response is 2; and "nearly every day" response is 3. Higher scores represents more depressive symptoms.
Change in quality of life measured by Euroqol, EQ-5D | Baseline, immediately after treatment completion, 1-month, 6-month and 12-month post-treatment
  Change in overall health from baseline to post treatment and follow up . EQ-5D is a standardized self-report measure of overall health status measured in terms of five dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using a three-level scale: 1 having no problems, 2 having some problems and 3 having extreme problems. A higher score indicate worse severity.
Change in Assessing Quality of Life 6 Dimensions (AQoL-6D) | Baseline, immediately after treatment completion, 1-month, 6-month and 12-month post-treatment
  Used to assess cost-effectiveness. 20 questions that assess different aspects of quality of life. The AQoL provides a utility score that ranges from 1.00 (full health) to 0.00 (death-equivalent health states) to -0.04 (health states worse than death).
Adverse events related to treatment measured by the Negative effects questionnaire | Immediately after treatment completion, 1-month, 6-month and 12-month post-treatment
  Self-rated questionnaire on negative effects. It contains 32 items that are scored on a five point Likert-scale (0-4) and differentiates between negative effects that are attributed to treatment and those possibly caused by other circumstances. The total score of the NEQ ranges from 0 to 80 points, a higher score reflects more negative effects.
Adverse events | Each treatment session and assessment point through study completion up to the 12-month follow up.
  Open ended question about recurrence of any adverse event
Change in Treatment Inventory of Costs in Psychiatric Patients (TIC-P) | Baseline, immediately after treatment completion, 1-month, 6-month and 12-month post-treatment
  Self-rated questionnaire on healthcare utilization and productivity losses in patients with a psychiatric disorder. The TIC-P questionnaire measures costs in two dimensions: use of health resources and loss of productivity. Lower cost is better.
Participants satisfaction with treatment, assessed by The Client Satisfaction Questionnaire (CSQ-8). | Immediately after treatment completion
  The CSQ-8 yields a single score measuring a single dimension of overall satisfaction. An "overall score" is calculated by summing the score on each of the eight scale item. Scores range from 8 to 32, with higher values indicating higher satisfaction.
Number of drop-outs from treatment and assessment | Baseline up to the 12-month follow up.
  Number of drop outs from treatment and assessment points will be calculated in each arm.

OTHER OUTCOMES:
Differences in treatment credibility between arms | Immediately after the first treatment session
  Measures treatment expectancy and rationale credibility. The CEQ is a 5-item measure of the treatment's credibility and the patients' expectations. The patients assess each domain on a 11-point likert scale (scored 0-10), with a total score ranging between 0-50 where higher score indicates higher credibility and higher expectations.
Differences in experience of working alliance between arms | Immediately after the third treatment session
  Measures the therapeutic alliance in therapy. The WAI-SR is a 12-item measure of the patient's experience of their working alliance with the therapist. The patients assess each item on a 7-point likert scale (scored 0-6), with a total score ranging between 0-72 where higher score indicates higher better working alliance according to the patient.
Adherence to treatment measured by the Therapist Adherence and Competence Rating Scale for prolonged exposure | Gold standard PE: Each treatment session up to week 15. Intensive PE: Each treatment session up to week 5
  The Therapist Adherence and Competence Rating Scale for prolonged exposure is a tool for measuring therapist adherence to treatment. The higher score, the higher adherence.
Change in emotional responding measured by the Subjective Distress Scale | Gold standard PE: Each treatment session up to week 15. Intensive PE: Each treatment session up to week 5
  Subjective level of distress will be measured using the Subjective units of distress (SUD) scale from 0-100. A higher score means higher distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Traumaprogrammet, Psykiatri Sydväst, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bragesjo M, Fina B, Ivanova E, Ivanov VZ, Ruck C. Study protocol for a single-blind, parallel-group, randomized, controlled superiority trial of intensive versus weekly delivered prolonged exposure for adults with post-traumatic stress disorder. Trials. 2024 Jun 12;25(1):381. doi: 10.1186/s13063-024-08218-2. PMID 38867309